CLINICAL TRIAL: NCT05645146
Title: Enhancing Long-Term Smoking Abstinence Among Cervical Cancer Survivors (Project ACCESS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MCC-21885
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Smoking Cessation; Cervical Cancer; High Grade Cervical Dysplasia
MeSH Terms: conditions — Smoking Cessation; Uterine Cervical Neoplasms | interventions — Tobacco Use Cessation Devices; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Standard Treatment (Active Comparator): Participants will receive a connection to the Tobacco Free Florida Quitline and a 12 week supply of nicotine replacement therapy (the patch and lozenges)
  Interventions: Behavioral: Smoking Cessation treatment delivered by Tobacco Free Florida Quitline; Drug: Nicotine patch; Drug: Nicotine Lozenge
- Group 2: Motivation and Problem Solving (MAPS) counseling (Experimental): Participants will receive a 12 week supply of nicotine replacement therapy (the patch and lozenges) along with the MAPS intervention, which consists of 6 MAPS counseling calls over 12 months, and individually tailored SMS text content driven by monthly smartphone delivered check-ins for 24 months
  Interventions: Drug: Nicotine patch; Drug: Nicotine Lozenge; Behavioral: Motivation and Problem Solving (MAPS) intervention

INTERVENTIONS:
Behavioral: Smoking Cessation treatment delivered by Tobacco Free Florida Quitline — Phone counseling with the state tobacco quitline
  Arms: Group 1: Standard Treatment
Drug: Nicotine patch — Participants will be provided with a 12 week supply of nicotine patches
Drug: Nicotine Lozenge — Participants will be provided with a 12 week supply of nicotine lozenges
Behavioral: Motivation and Problem Solving (MAPS) intervention — MAPS is a phone counseling approach to facilitating smoking cessation among cervical cancer survivors, which uses a combined motivational interviewing and social cognitive theory based approach to smoking cessation. Participants will receive 6 MAPS based counseling calls over 12 months, along with personally-tailored SMS-delivered text based messages delivered to the participants phone over 2 years.
  Arms: Group 2: Motivation and Problem Solving (MAPS) counseling

SUMMARY:
The goal of this research study is to compare the efficacy of a treatment approach that comprises both Motivation And Problem-Solving (MAPS)-based telephone counseling and a personally-tailored SMS-delivered text-based approach to quitline-delivered smoking cessation treatment to help participants with a history of cervical cancer or high-grade cervical dysplasia quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* At least 100 cigarettes or more smoked in participants lifetime
* Speaks English
* Currently smoke 1 cigarette or more in the past 30 days
* History of cervical cancer or high grade cervical dysplasia
* Has a working smartphone
* Has a valid home address
* Reside in Florida at the time of study enrollment

Exclusion Criteria:

* Receiving behavioral or pharmacological tobacco treatment
* Household member enrolled in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — cervical cancer or cervical dysplasia patients
Enrollment: 360 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
MAPS vs Standard Treatment in facilitating long term smoking abstinence | at 24 months
  The primary outcome of this study is self-reported, 7 day point prevalence abstinence over time through the 24 month assessment where participants who report no smoking in the previous 7 days at follow-up assessment are considered abstinent.
  Efficacy of MAPS vs Standard Treatment will be measured by comparing the number of participants in each group who were able to quit smoking and maintain smoking abstinence for 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Vidrine, PhD, MS, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- [Derived] Vidrine JI, Fennell BS, Simmons VN, Sutton SK, Jones SR, Woodward HW, Hoogland CE, Vidrine DJ. Enhancing long-term smoking abstinence among individuals with a history of cervical intraepithelial neoplasia or cervical cancer (Project ACCESS): protocol for a randomized clinical trial. BMC Public Health. 2023 Jul 4;23(1):1284. doi: 10.1186/s12889-023-16189-3. PMID 37403057